CLINICAL TRIAL: NCT03790098
Title: Can Yoga Decrease Pain and Inflammation Among Women Aged 60 or Older: A Pilot Feasibility Study
Brief Title: Flow-Restorative Yoga to Decrease Pain and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1809008271
Record Dates: First submitted 2018-12-19; First posted 2018-12-31 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Pain; Inflammation
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Intervention Model Description: Group 1 Participants attend Restorative-Flow Yoga classes, two times per week with a certified yoga instructor and have at-home supplemental materials. Group 2 receive the at-home supplemental materials after outcome visit corresponding to after the 24 classes.
Masking Description: Randomization to arm follows the baseline assessment visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Class Participants (Experimental): Group 1 participants will meet twice per week for one hour to practice restorative-flow yoga with a certified yoga instructor. There will be a total of 24 classes. Group 1 participants will also receive an at-home supplemental booklet, a yoga video led by the class instructor, and encouragement to practice two additional days each week at home. They will be asked to fill out a form to record their at-home practice.
  Interventions: Behavioral: Restorative-Flow Yoga
- No Classes (No Intervention): Group 2 participants will not attend yoga classes as part of the study and will be asked not to begin yoga classes outside the study. After the 24 classes, they will be given the 'at-home' supplemental materials.

INTERVENTIONS:
Behavioral: Restorative-Flow Yoga — Restorative yoga consists of a series of gentle poses, supported by props, with an emphasis on breathing and relaxing; as opposed to stretching or contracting muscles, it is designed to support muscles. Flow yoga consists of a series of linked poses synchronized with the breath.
  Arms: Yoga Class Participants

SUMMARY:
The Restorative Flow Yoga Study is a pilot project looking at whether restorative flow yoga will reduce inflammation and pain in women 60 and older who experience chronic pain.

DETAILED DESCRIPTION:
The aims of the study are to (1) evaluate the feasibility of implementing a restorative-flow yoga randomized trial (24 classes, held twice per week) for women aged 60 or older who experience chronic pain; and (2) evaluate the preliminary efficacy of restorative-flow yoga to decrease pain and inflammation among women aged 60 or older. Feasibility measures will include three areas of focus (a) acceptability, (b) implementation, and (c) demand and use, evaluated using recruitment rate, retention rate, class and home practice adherence rates, resource utilization, and safety. With a sample size of 40, this pilot feasibility study is likely under-powered to determine intervention effects. However, the study will evaluate preliminary efficacy of the yoga intervention. The study will measure BMI, blood pressure, resting heart rate, physical function measures, and inflammatory markers C-reactive protein, IL-2, IL-1β, TNF-α, IL-6, IL-4, and IL-10) at baseline and outcome assessments (after 24 class sequence).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 60 or older
* Report AVERAGE severity of 3 or higher on the brief pain inventory
* Blood pressure is less than 160/100 mm Hg
* Heart rate is between 55-110 bpm
* Able and willing to obtain physician's approval to participate

Exclusion Criteria:

* Currently practicing yoga two or more times per week
* Cognitively impaired

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-04-27 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in inflammatory markers | Baseline and outcome (after 24 class sequence, about 14 weeks)
  Change from baseline measures of C-reactive protein, IL-2, IL-1β, TNF-α, IL-6, IL-4, and IL-10
Change from baseline in Average Pain on The Brief Pain Inventory | Baseline and outcome (after 24 class sequence, about 14 weeks)
  Change from baseline self-report of AVERAGE pain on the severity scale of the The Brief Pain Inventory (BPI) where where 0=no pain and 10=pain as bad as you can imagine. The BPI is a widely used measurement tool for assessing clinical pain.

SECONDARY OUTCOMES:
Change from baseline in the 'Chair Stand Test' | Baseline and outcome (after 24 class sequence, about 14 weeks)
  The 'Chair Stand Test' is a count of the number of full stands that can be completed in 30 seconds with arms folded across chest. It is one of six functional fitness/ senior fitness tests that will be measured at baseline and outcome to assess change from baseline.
Change from baseline in the 'Arm Curl Test' | Baseline and outcome (after 24 class sequence, about 14 weeks)
  The 'Arm Curl Test' is a count of the number of bicep curls that can be completed in 30 seconds holding a hand weight of 5 lbs. for women. It is one of six functional fitness/ senior fitness tests that will be measured at baseline and outcome to assess change from baseline.
Change from baseline in the '2-Minute Step Test' | Baseline and outcome (after 24 class sequence, about 14 weeks)
  The '2-Minute Step Test' is a count of the number of full steps completed in 2 minutes, raising each knee to a point midway between the kneecap and hip bone. It is one of six functional fitness/ senior fitness tests that will be measured at baseline and outcome to assess change from baseline.
Change from baseline in the 'Chair Sit-and-Reach Test' | Baseline and outcome (after 24 class sequence, about 14 weeks)
  The 'Chair Sit-and-Reach Test' is a measure of the distance that a participant can reach toward or past her toes when stretching forward from a seated position. It is one of six functional fitness/ senior fitness tests that will be measured at baseline and outcome to assess change from baseline.
Change from baseline in the 'Back Scratch Test' | Baseline and outcome (after 24 class sequence, about 14 weeks)
  The 'Back Scratch Test' is a measure of the distance or overlap between her fingers, as a participant reaches behind her back. It is one of six functional fitness/ senior fitness tests that will be measured at baseline and outcome to assess change from baseline.
Change from baseline in the '8-foot up and go' | Baseline and outcome (after 24 class sequence, about 14 weeks)
  The '8-foot up and go' is measure of the number of seconds required to get up from a seated position, walk 8 feet, turn, and return to seated position. It is one of six functional fitness/ senior fitness tests that will be measured at baseline and outcome to assess change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Seguin, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seguin-Fowler R, Graham M, Ward J, Eldridge G, Sriram U, Fine D. Feasibility of a yoga intervention to decrease pain in older women: a randomized controlled pilot study. BMC Geriatr. 2020 Oct 12;20(1):400. doi: 10.1186/s12877-020-01818-y. PMID 33046009